CLINICAL TRIAL: NCT06429709
Title: Utility of Advanced Ultrasound Otoscope In The Diagnosis of Acute Otitis Media
Brief Title: Utility of Advanced Ultrasound Otoscope In The Diagnosis of AOM
Status: Active, not recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: OtoNexus Medical Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Yi-Chun Carol Liu, Associate Professor, Baylor College of Medicine
Other Study IDs: H-50018
Record Dates: First submitted 2024-04-16; First posted 2024-05-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-05

CONDITIONS: Otitis Media Recurrent; Middle Ear Infection; Ear Infection
Keywords: Otoscope; Tympanogram; Effusion; Ultrasound
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Algorithm Development: Ultrasound and signal information and visual otoscopic images will be collected with an engineering prototype otoscope device for children scheduled for tympanostomy tube surgery. Images of each of the child's ears will be taken by the advanced ultrasound otoscope device. Data collected will include ear laterality, surgical and lab findings of the effusion (present or absent) and characteristics as reported by the surgeon. The middle ear fluid which is usually suctioned will be collected in a trap chamber- Tympap- and this collected fluid will be send for analysis to microbiology. The pathology results will be recorded to correlate ultrasound signals to surgical findings
  Interventions: Device: Advanced Ultrasound Otoscope
- Clinical Validation: The clinical validation phase includes the same procedures as the algorithm development phase only, the clinical validation phase is a double blind study where ultrasound score is compared to surgical findings and lab analysis.
  Interventions: Device: Advanced Ultrasound Otoscope

INTERVENTIONS:
Device: Advanced Ultrasound Otoscope — The Advanced Ultrasound Otoscope is a tool for visualization of the human tympanic membrane and detection of middle ear effusion type

SUMMARY:
The objective of this study is to collect ultrasound signal information and visual otoscopic images with an engineering prototype device for children scheduled for tympanostomy tube surgery for the purpose of algorithm development.

DETAILED DESCRIPTION:
The objective of this study is to collect ultrasound signal information and visual otoscopic images with an engineering prototype device for children scheduled for tympanostomy tube surgery for the purpose of algorithm development.

After informed consent from a parent or guardian is obtained, ultrasound and visual data will be collected for each of the child's ears. The images will be taken with the Advanced Ultrasound Otoscope device. The ear laterality will be noted as well as any infection present in the fluid, non-infected fluid, or normal findings in the middle ear as reported by the surgeon. No identifiable data will be recorded. Each study participant will be given a unique study number that will be linked to the images and middle ear findings. No additional information is gathered including age, sex, name or other PHI. The images and corresponding study data will be stored on a password protected smartphone or tablet as well as on a password protected external hard drive. Other characteristics that will be collected include surgical and lab findings regarding effusion, presence or absence (i.e. effusion). The middle ear fluid which is usually suctioned will be collected in a trap chamber- Tympap- and this collected fluid will be sent to the microbiology laboratory for analysis

Investigators will be collecting ultrasound and visual data from the tympanic membrane. The images the investigators are collecting are optical images of the surface of the tympanic membrane. The waveforms do not traverse the body tissue, the tympanic membrane is a strong reflector, and the signal is returned to the ultrasound transducer for processing the waveform from an analog to a digital signal. The power of the ultrasound signal is 1/1000th of the ultrasound power used for fetal imaging which is considered safe.

ELIGIBILITY:
Inclusion Criteria:

* Newborn to 12 years of age
* Receiving first set of pressure equalization (PE) tubes, even if coordinated with other procedures such as adenoidectomy
* Indication for surgery includes recurrent acute otitis media, chronic otitis media with effusion, Eustachian tube dysfunction, and/or hearing loss.

Exclusion Criteria:

* Cholesteatoma, tympanic membrane perforation, myringitis
* History of PE tube placement or PE tubes currently in place.

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators will be recruiting patients between 0 months and 12 years of age who meet the listed inclusion criteria and do not meet any of the listed exclusion criteria. The investigators are not selecting patients based on race/ethnicity or gender/sex. Parents must be fluent in either English or Spanish.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Device Performance | 2 years and 6 months
  Correlations of device measurements and ultrasound data for Noninfected fluid and Bacterial Fluid to the gold standard of surgeon's findings at myringotomy.

SECONDARY OUTCOMES:
Device Usability | 1 year
  Evaluate the usability of the Advanced Ultrasound Otoscope device in pediatric patients as measured by the ability of the device to fit in subjects' external auditory canals and obtain a tympanic mobility measurement(s).

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Raynor, MD, Study Chair — Baylor College of Medicine; Yi-Chun Liu, MD, Principal Investigator — Baylor College of Medicine; Shraddha Mukerji, MD, Study Chair — Baylor College of Medicine; Jennifer Yan, MD, Study Chair — Baylor College of Medicine; Sonal Saraiya, MD, Study Chair — Baylor College of Medicine; Mary E Williamson, MD, Study Chair — Baylor College of Medicine; Henri Traboulsi, MD, Study Chair — Baylor College of Medicine; Anna Messner, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No